CLINICAL TRIAL: NCT02254941
Title: Observational Study to Evaluate the Use of Targeted Therapies in Metastatic Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Grupo Espanol Multidisciplinario del Cancer Digestivo (Other)
Responsible Party: Sponsor
Other Study IDs: GEMCAD 1401
Record Dates: First submitted 2014-09-23; First posted 2014-10-02 (Estimated); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Metastatic Colon Cancer
Keywords: Metastatic Colon Cancer; Monoclonal antibodies; Chemotherapy; First line
MeSH Terms: conditions — Colonic Neoplasms | interventions — Drug Therapy; Antibodies, Monoclonal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Colon biopsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Active comparator: Chemotherapy: Metastatic colon cancer and first line treatment with conventional chemotherapy without monoclonal antibody.
  Interventions: Drug: Chemotherapy
- Experimental: Chemotherapy plus mAb: Metastatic colon cancer and first line treatment with conventional chemotherapy plus monoclonal antibody
  Interventions: Biological: Chemotherapy plus monoclonal antibody

INTERVENTIONS:
Drug: Chemotherapy — Metastatic colon cancer, first line treatment with conventional chemotherapy
  Other Names: Standard Chemotherapy
  Groups: Active comparator: Chemotherapy
Biological: Chemotherapy plus monoclonal antibody — Metastatic colon cancer, first line treatment with conventional chemotherapy plus monoclonal antibody
  Other Names: Standard CHemotherapy plus monoclonal antibody
  Groups: Experimental: Chemotherapy plus mAb

SUMMARY:
The purpose of this study is to evaluate, in terms of overall survival, the benefit of monoclonal antibodies in the start time of the diagnosis of advanced disease or administer a deferred basis after progression to treatment with chemotherapy alone. Initially expected target population was 1950 patients (pts), in 2015 protocol was ammended to 1028 patients, because the size was sufficient to evaluate the superiority of the use of monoclonal antibodies the start time of the diagnosis against deferred use, with HR of 0.8, power of 90% and an alpha of 0.05. Finally in July 2018, recruitment was completed with a total of 1104 patients enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with metastatic colorectal cancer with biopsy positive for adenocarcinoma.
* ECOG PS0-2.
* Who have not received prior chemotherapy treatment for metastatic disease.
* Measurable or evaluable disease.
* No previous surgery for metastatic disease. Surgery for metastasis allowed after inclusion in the study aftercare at the discretion of investigadors.
* Chemotherapy treatment with doublets (CAPOX, FOLFOX, FOLFIRI)

Exclusion Criteria:

* Patients older than 70 years with frailty criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Metastatic colorectal cancer. Adenocarcinoma. First line treatment
Sampling Method: Non-Probability Sample
Enrollment: 1104 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From July 2018 (LPI), 24 months
  From date of inclusion until the date of death from any cause.

SECONDARY OUTCOMES:
Validate prognostic score GEMCAD | From August 2014, up to 36 months
  The two main prognostic scores for metastatic colorectal cancer (Kohne and GERCOR) do not account for resectability of liver-only metastasis (LiM) and thus are limited as treatment guidance. We propose a classification of patients based on LiM resectability, performance status (PS) and lactate dehydrogenase (LDH) levels and compare its discrimination capacity against Kohne and GERCOR scores.
  GEMCAD score: patients are classified as stage 1 if LiM are considered resectable (<4 nodules and <5 cm diameter) or potentially resectable (>4 and <10 nodules or >5 cm diameter), PS 0-1 and LDH < 1.5 ULN; stage 2 if LiM are not resectable or with extrahepatic spread, PS 0-1 and LDH < 1.5 ULN; stage3 if PS 2 or LDH > 1.5 ULN.
  This score, Kohne, and GERCOR scores will be tested for discrimination using Harrel's C index (HCI, higher is better) and calibration using Akaike information criterion (AIC, smaller is better) of progression-free survival (PFS) and overall survival (OS).
To compare GERCOR and Köhne classification with GEMCAD classification | From August 2014, up to 36 months
  The two main prognostic scores for metastatic colorectal cancer (Kohne and GERCOR) do not account for resectability of liver-only metastasis (LiM) and thus are limited as treatment guidance. We propose a classification of patients based on LiM resectability, performance status (PS) and lactate dehydrogenase (LDH) levels and compare its discrimination capacity against Kohne and GERCOR scores.
  This score, Kohne, and GERCOR scores will be tested for discrimination using Harrel's C index (HCI, higher is better) and calibration using Akaike information criterion (AIC, smaller is better) of progression-free survival (PFS) and overall survival (OS).
Evaluate Sadananda cellular phenotype classification | From August 2014, up to 36 months
Study other variables to identify whether there is group of patients who may benefit from monoclonal antibodies for the treatment of first-line chemotherapy | From August 2014, up to 36 months
  Study whether there are demographic variables, analytical or related tumor and its extension to allow us to identify whether there is group of patients who may benefit from monoclonal antibodies for the treatment of first-line chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Joan Maurel, MD PhD, Study Chair — Hospital Clinic of Barcelona
Locations (48):
- Spain (48):
  - Hospital Virgen de los Lirios, Alcoy, Alicante
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Universitario del Vinalopó, Elche, Alicante
  - Hospital General Universitario de Elda, Elda, Alicante
  - Hospital Universitario de Torrevieja, Torrevieja, Alicante
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza, Aragon
  - Hospital Granollers, Granollers, Barcelona
  - Corporació Sanitària Parc Taulí, Sabadell, Barcelona
  - Hospital General de Catalunya, Sant Cugat del Vallès, Barcelona
  - Hospital de Terrasa, Terrassa, Barcelona
  - Hospital General de Vic, Vic, Barcelona
  - Hospital Universitario Virgen del Puerto de Plasencia, Plasencia, Cáceres
  - Hospital de Donostia, San Sebastián, Guipúzcoa
  - Centro Oncologico de Galicia, A Coruña, La Coruña
  - Hospital Universitario de Gran Canaria Doctor Negrín, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Puerta de Hierro de Majadahonda, Majadahonda, Madrid
  - Hospital Son Espases, Palma, Malllorca
  - Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Costa del Sol, Marbella, Málaga
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Hospital Lluis Alcanyis de Xátiva, Xàtiva, Valencia
  - Hospital Obispo Polanco, Teruel, Zaragoza
  - Hospital Infanta Cristina de Badajoz, Badajoz
  - Centre Mèdic Teknon, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hosptial de l'Esperit Sant de Barcelona, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital Plató, Barcelona
  - Hospital Universitari Sagrat Cor, Barcelona
  - Consorcio Hospitalario Provincial de Castellón, Castelló
  - Hospital San Pedro de Alcantara Cáceres, Cáceres
  - Hospital General de Ciudad Real, Ciudad Real
  - Hospital Univeritari Dr. Josep Trueta, Girona
  - Hospital Arnau de Vilanova de Lleida, Lleida
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital La Paz, Madrid
  - Hospital Althaia, Manresa
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Morales Meseguer, Murcia
  - Complejo Hospitalario Universitario de Ourense, Ourense
  - Hospital Universitari Son Llàtzer, Palma de Mallorca
  - Hospital Provincial de Pontevedra, Pontevedra
  - Hospital de Sagunto, Sagunto
  - Instituto Valenciano de Oncologia, Valencia
  - Hospital Doctor Peset, Valencia
  - Hospital Universitario y Politécnico de La Fe, Valencia
  - Complejo Hospitalario Universitario de Vigo, Vigo
  - Hospital Miguel Servet, Zaragoza